CLINICAL TRIAL: NCT04536025
Title: Shared Decision Making Aid for Prosthetic Design
Acronym: D-MAP
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Orthotic and Prosthetic Education and Research Foundation (OPERF) (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1070
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Amputation; Prosthesis User
Keywords: Lower Limb Amputation; Decision Making

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prosthetists: Up to 24 prosthetists who are actively providing prosthetic care to people with lower limb amputation will be recruited for participating in focus groups to describe their decisional needs for providing prostheses to people with lower limb amputation.
  Interventions: Other: Qualitative focus group interviews
- People with lower limb amputation: An estimated 14 people within 1 year from lower limb amputation, receiving their first prosthesis will be recruited for individual semi-structured interviews to describe their decisional needs for provision of a prosthesis.
  Interventions: Other: Qualitative semi-structured interviews
- Expert working group: The expert working group will consist of at least 5 and up to 12 people with LLA actively receiving prosthetic care, and at least 5 and up to 12 prosthetic care providers with greater than 5 years of experience. Individuals will be invited to join the expert working group based on expertise, and representation of key stakeholders relevant to the prosthetic design process.
  Interventions: Other: Qualitative focus group interviews; Other: Qualitative semi-structured interviews

INTERVENTIONS:
Other: Qualitative focus group interviews — Prosthetists and/or expert working group members will participate in qualitative focus group interviews up to 120 minutes in length.
  Groups: Expert working group; Prosthetists
Other: Qualitative semi-structured interviews — People with lower limb amputation and/or expert working group members will participate in qualitative individual, semi-structured interviews approximately 60 minutes in length.
  Groups: Expert working group; People with lower limb amputation

SUMMARY:
This study is designed to learn more about decision making for prosthetic design, with the goal of producing a decision making aid for prosthetic design decisions.

DETAILED DESCRIPTION:
The overarching hypothesis of this work is that the lack of shared decision making (SDM) for prosthetic design and failure to match patient expectations with a prosthetic design plan result in poor health outcomes for patients with LLA. Shared decision making (SDM) is where clinicians and patients share the best available evidence for comparing options in order to achieve informed preferences for making health decisions. A patient's involvement in their health care process is known to affect their satisfaction, adherence to care programs, and health outcomes. Clinical decision aids (DAs) support patients in SDM and making informed health decisions, by providing information on the available options and associated outcomes. DAs are intended to help patients clarify their values associated with the options and potential outcomes, to create a platform for communication with healthcare providers. DAs have been shown to improve patient knowledge and realistic expectations for given health options. This project aims to examine how to better align patient and clinician values and expectations by developing a DA for prosthetic design decision options, to support SDM between patients receiving their first prosthesis and prosthetic care providers. This proposal will be guided by the International Patient Decision Aids Standards (IPDAS).

Aim 1: Qualitatively define the key determinants and decisional needs of new prosthetic patients (n=14) and prosthetic care providers (n=20- 24) during prosthetic design, via semi structured interviews with patient participants and focus groups with prosthetist participants.

Expected Result 1.1: Key determinants and decisional needs for prosthetic design will be defined using content analysis guided by the Ottawa Decision Support framework9 for patients making health decisions, and the Model for Shared Decision Making in Clinical Practice.

Expected Result 1.2: Key stakeholders who contribute directly to prosthetic design decisions (e.g., patients with LLA, prosthetists, physicians, caregivers, close friends or family members) will be identified via purposive sampling, to inform the target end users of a DA prototype.

Aim 2: Synthesize the evidence for prosthetic design decision options to develop a DA prototype.

Expected Result 2.1: Via systematic literature review, a DA prototype will be developed from the evidence on prosthetic design decision options associated with decisional needs identified in Aim 1.

Aim 3: Assess the DA prototype's accuracy, comprehensibility, and usability through alpha testing with an expert working group of patients with LLA and prosthetic care providers.

Expected Result 3.1: Quantitative results from a Likert scale measurement of the DA prototype's accuracy, comprehensibility and usability will inform revisions to the DA prior to use in a pilot clinical trial.

Expected Result 3.2: Qualitative feedback on the DA prototype's accuracy, comprehensibility, and usability will inform directed iterative revision for the DA prototype and implementation methods for use in a pilot clinical trial.

ELIGIBILITY:
Group 1 Prosthetist Inclusion Criteria:

* At least 18 years of age
* Prosthetists actively providing prosthetic care to people with lower limb amputation

Group 1 Prosthetist Exclusion Criteria:

* Unable to participate in a 1 hour phone or video conference
* Non-English speaking

Group 2 Patient Inclusion Criteria:

* At least 18 years of age
* People who have a lower limb amputation
* People within 1 year since their first amputation
* Amputation levels ranging between above the ankle and below the hip

Group 2 Patient Exclusion Criteria:

* Unable to participate in a 1 hour phone or video conference
* Non-English speaking

Group 3 Expert Working Group Inclusion Criteria:

* At least 18 years of age
* People who have a lower limb amputation ranging between above the ankle and below the hip *OR* Prosthetists with at least 5 years experience providing prosthetic care to people with lower limb amputation.

Group Expert Working Group Exclusion Criteria:

* Unable to participate in a 1 hour phone or video conference
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited for three groups:
  1. Prosthetists who actively provide prosthetic care, for focus group qualitative interviews to determine decisional needs for prosthetic decisions.
  2. People with lower limb amputation who are within their first year after amputation and using their first prosthesis, for individual semi-structured qualitative interviews to determine decisional needs for prosthetic decisions.
  3. An Expert Working Group of patients with lower limb amputation and prosthetists, for collecting data on the comprehensibility, usability, and acceptability of the Decision Aid Prototype. Prosthetists will have at least 5 years of experience providing prosthetic care, and patients with lower limb amputation will be actively receiving prosthetic care.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory L Christiansen, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
Started | 38 | 17 | 11
Completed | 38 | 17 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prosthetists: Qualitative Focus Groups
- People With Lower Limb Amputation: Qualitative Individual Interviews
- Expert Working Group: Qualitative Focus Groups, Individual Interviews, Quantitative Surveys
- Total: Total of all reporting groups
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group | Total
Number analyzed (Participants) | 38 | 17 | 11 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 13 | 8 | 59
  >=65 years | 0 | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 6 | 23
  Male | 28 | 10 | 5 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 36 | 15 | 11 | 62
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 35 | 14 | 10 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 17 | 11 | 66
Qualitative Focus Groups [Count of Participants; unit: Participants] — All study participants participated in either qualitative focus groups or qualitative semi-structured individual interviews. A semi-structured interview guide was utilized, and interviews were transcribed and qualitatively analyzed using directed content analysis.
  Participants | 38 | 17 | 11 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Participated in and Completed 1 Hour Qualitative Interview Data Collection Via a Semi Structured Interview Guides
Description: During 1 hour semi structured interviews with participants, questions about the decisional needs of patients and prosthetists for Prosthetic Design Decisions were asked. Because qualitative data is not numerical, the transcripts of each interview were analyzed using directed content analysis using the Ottawa Decision Support Framework, and the Elwyn Shared Decision Making Model, and resulting final qualitative themes were used to guide the content in the development of a decision aid for prosthetic design. Qualitative data is not numerical, and only the number of participants who complete the semi structured interviews was able to be numerically recorded and analyzed.
Time Frame: Data collection of the semi structured qualitative interview occurred at the baseline time point only, lasting an average of 1 hour during 1 day.
Measure: Count of Participants; unit: Participants
Groups:
- Prosthetists: 38 prosthetists who are actively providing prosthetic care to people with lower limb amputation were recruited for participating in focus groups to describe their decisional needs for providing prostheses to people with lower limb amputation.
  Qualitative focus group interviews: Prosthetists and/or expert working group members will participate in qualitative focus group interviews up to 120 minutes in length.
- People With Lower Limb Amputation: 17 people within 1 year from lower limb amputation, receiving their first prosthesis were recruited for individual semi-structured interviews to describe their decisional needs for provision of a prosthesis.
  Qualitative semi-structured interviews: People with lower limb amputation and/or expert working group members will participate in qualitative individual, semi-structured interviews approximately 60 minutes in length.
- Expert Working Group: The expert working group consisted of 6 people with LLA actively receiving prosthetic care, and 5 prosthetic care providers with greater than 5 years of experience. Individuals were invited to join the expert working group based on expertise, and representation of key stakeholders relevant to the prosthetic design process.
  Qualitative focus group interviews: Prosthetists and/or expert working group members participated in qualitative focus group interviews up to 120 minutes in length.
  Qualitative semi-structured interviews: People with lower limb amputation and/or expert working group members participated in qualitative individual, semi-structured interviews approximately 60 minutes in length.
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
Number analyzed (Participants) | 38 | 17 | 11
Participants | 38 | 17 | 11

2. Primary Outcome: Accuracy of the Decision Aid Prototype, as Measured in Percentage.
Description: The Accuracy of the Decision Aid is a single item Likert scale measure of the degree to which the decision aid's revised content, advantages, and disadvantages in the decision aid aligns with the scientific evidence available on the prosthesis design decision outcomes. This scale includes 1 question, with a range of response scoring from 1 to 5. 1 represents low accuracy of the decision aid, while 5 represents high accuracy of the decision aid. The final score is converted to a percentage for all respondents (ranging 0% to 100%, with a higher percentage representing greater accuracy).
Time Frame: Data collection occurred at the baseline time point only, lasting an average of 1 hour during 1 day.
Population: Accuracy was only evaluated in the Expert Working Group
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
Number analyzed (Participants) | 0 | 0 | 10
percentage |  |  | 96.0 (5.2)

3. Primary Outcome: Comprehensibility of the Decision Aid Prototype, as Measured by a Likert Scale
Description: The Comprehensibility of the Decision Aid is a single item Likert scale measure of the degree to which the information in the Decision Aid was understandable and covers information necessary for making an informed decision about prosthesis design. This scale includes 1 question, with a range of response scoring from 1 to 5. 1 represents low comprehensibility of the decision aid, while 5 represents high comprehensibility of the decision aid. The final score is calculated as a percentage (ranging 0% to 100%, with a higher percentage representing greater comprehensibility) for all participants.
Time Frame: Data collection occurred at the baseline time point only, lasting an average of 1 hour during 1 day.
Population: Only the Expert Working Group participated in Comprehensibility survey data collection.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
Number analyzed (Participants) | 0 | 0 | 10
percentage |  |  | 96.0 (7.0)

4. Primary Outcome: Usability of the Decision Decision Aid Prototype, as Measured by a Likert Scale
Description: The Usability of the Decision Aid is a single item Likert scale measure of the degree to which the Decision Aid prototype was acceptable, clear, understandable, and effective in use. This scale includes 1 question, with a range of response scoring from 1 to 5. 1 represents low usability of the decision aid, while 5 represents high usability of the decision aid. The final score is calculated as a percentage for all respondents (ranging 0% to 100%, with a higher percentage representing greater usability).
Time Frame: Data collection occurred at the baseline time point only, lasting an average of 1 hour during 1 day.
Population: Only Expert Working Group Members participated in Usability Survey Data collection.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
Number analyzed (Participants) | 0 | 0 | 10
percentage |  |  | 93.0 (8.2)

5. Secondary Outcome: Participant Preferences for Personal Preference Towards Control in a Health Decision, as Measured by the Control Preferences Scale Survey
Description: The control preference scale is a measure of the degree of control an individual wants to assume when decisions are being made about medical treatment. This scale was adapted to this study, to include 5 questions with a range of response scores from 1 to 5 for each question (totaling a final score ranging from 5 to 25). 1 the degree of control an individual wants to assume when decisions are being made about medical treatment represents a more passive provider controlled preference for making a decision, while 5 represents a more active patient controlled preference for making a decision.
Time Frame: Data collection occurred at the baseline time point only, lasting an average of 1 hour during 1 day.
Population: Data from the Control Preference Scale was only collected and analyzed in the Prosthetists group and the People with Lower Limb Amputation Group, not the Expert Working Group.
Measure: Mean (Standard Deviation); unit: units on a scale, range 5-25
Groups:
- Prosthetists: 38 prosthetists who are actively providing prosthetic care to people with lower limb amputation.
- People With Lower Limb Amputation: 17 people within 1 year from lower limb amputation, receiving their first prosthesis.
- Expert Working Group: The expert working group consisted of 6 people with LLA actively receiving prosthetic care, and 5 prosthetic care providers with greater than 5 years of experience. Individuals were invited to join the expert working group based on expertise, and representation of key stakeholders relevant to the prosthetic design process.
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
Number analyzed (Participants) | 38 | 17 | 0
units on a scale, range 5-25 | 15.5 (2.1) | 15.4 (4.5) |

6. Secondary Outcome: Perceived Ability to Find and Use Health Information, Via the eHealth Literacy Scale Survey
Description: The eHealth Literacy scale survey is a 10-item measure of electronic Health literacy developed to measure patient's combined knowledge, comfort, and perceived skills at finding, evaluating, and applying electronic health information to health problems. This scale includes 10 questions with a range of response scores from 1 to 5 for each question (totaling a final score ranging from 10 to 50). 1 represents low electronic health literacy, while 5 represents higher electronic health literacy.
Time Frame: Data collection occurred at the baseline time point only, lasting an average of 1 hour during 1 day.
Population: Data from the eHealth Literacy Scale Survey was only collected from the Prosthetists group and the People with Lower Limb Amputation group, and was not collected from the Expert Working group
Measure: Mean (Standard Deviation); unit: units on a scale, range 10-50
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
Number analyzed (Participants) | 38 | 17 | 0
units on a scale, range 10-50 | 41.7 (4.1) | 36.3 (6.7) |

ADVERSE EVENTS:
Time Frame: Because all participants were seen at one time point (Data collection occurred at the baseline time point only, lasting an average of 1 hour during 1 day), All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored or assessed.
Description: Because all participants were seen at one time point (Data collection occurred at the baseline time point only, lasting an average of 1 hour during 1 day), All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored or assessed.
Arm/Group | Prosthetists | People With Lower Limb Amputation | Expert Working Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT04536025/Prot_SAP_000.pdf